CLINICAL TRIAL: NCT00928252
Title: Chemotherapy Response Monitoring With 18F-choline PET/CT in Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Queen's Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sandi Kwee, Sandi A. Kwee, M.D., Queen's Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RA-2008-069; R21CA139687 (NIH)
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Results first posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-07

CONDITIONS: Hormone Refractory Prostate Cancer
Keywords: Hormone Refractory Prostate Cancer; Castrate Resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Received 18F-fluorocholine PET/CT (Experimental): IV fluorine-18 labeled methylcholine before PET/CT
  Interventions: Drug: IV fluorine-18 labeled methylcholine before PET/CT

INTERVENTIONS:
Drug: IV fluorine-18 labeled methylcholine before PET/CT — Intervention at pre-treatment, and at two timepoints post treatment intiation.
  Other Names: 18F-fluorocholine PET/CT

SUMMARY:
The purpose of this study is to determine whether imaging with 18F-choline PET/CT can provide information that may help guide subsequent investigational or clinical treatments for patients with advanced (hormone-refractory) metastatic prostate cancer.

DETAILED DESCRIPTION:
Patients who meet eligibility criteria and are enrolled will undergo whole-body imaging with 18F-choline PET/CT at 3 time points during the course of treatment that is indicated for castrate resistant prostate cancer. The 1st PET/CT scan is performed at baseline before treatment initiation. The 2nd and 3rd scans are performed at two other treatment-releated timepoints or at approximately 1 month and 3 months after treatment initiation. Change in lesion 18F-choline uptake from baseline measured at each time point will be determined. Cancer 18F-choline uptake will be evaluated as a marker of therapeutic response in comparison to PSA response and symptom scores. Treatment-related changes in tumor 18F-choline uptake occur will be studied after the second and third PET scans to determine the acuity by which changes in tumor 18F-choline uptake can be expected following specific treatments for castrate-resistant prostate cancer. The study evaluates a diagnostic intervention and the treatments themselves are not considered part of the investigation. All treatment decisions will be made independent of the study and must be deemed clinically-warranted by a treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent.
2. Men, over 18 years of age, with histologically-confirmed diagnosis of prostate cancer
3. History of treatment by complete androgen blockade for greater than 3 months prior to enrollment
4. Progressive disease evidenced by 2 consecutive rises in PSA measured at least 1 week apart, with the absolute value of the latest PSA > 5.0 ng/ml.
5. A rise in PSA following anti-androgen drug withdrawal, above the last PSA value before withdrawal.
6. Patient has agreed to treatment for hormone-refractory (ie. castrate-resistant) prostate cancer under supervision of a medical oncologist, urologist, radiation oncologist or nuclear medicine physician. Treatments indicated for HRPC are docetaxel-, cabazitaxel-, or mitoxantrone-based chemotherapy, abiraterone, radium-223, enzalutamide, or sipulecuil-T.

Exclusion Criteria:

1. Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or superficial transitional cell carcinoma of the bladder.
2. Serious underlying medical conditions that would otherwise impair the patient's ability to undergo imaging.
3. Patient weighs over 350 lbs (due to scanner weight limit).
4. Clinical life expectancy < 12 weeks.
5. Participated in other radioactive drug studies where estimated total cumulative dose within 1 year is > 0.05 Sievert for whole body, active blood-forming organs, eye lens, gonads, or 0.15 Sievert for other organs.
6. Concurrent Therapy. Allowed: Prior or concurrent chemotherapy, but must be > 12 weeks since last treatment at enrollment; prior or concurrent hormonal therapy; prior surgery; prior or concurrent bisphosphonate; prior or concurrent receptor/biologic agent allowed if given on approved study protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandi A Kwee, MD, Principal Investigator — The Queen's Medical Center
Locations (1):
- The Queen's Medical Center, Honolulu, Hawaii, United States

REFERENCES:
- [Derived] Lee J, Sato MM, Coel MN, Lee KH, Kwee SA. Prediction of PSA Progression in Castration-Resistant Prostate Cancer Based on Treatment-Associated Change in Tumor Burden Quantified by 18F-Fluorocholine PET/CT. J Nucl Med. 2016 Jul;57(7):1058-64. doi: 10.2967/jnumed.115.169177. Epub 2016 Feb 16. PMID 26912444

RESULTS

PARTICIPANT FLOW:
Groups:
- Received 18F-fluorocholine PET/CT: 18F-fluoromethylcholine IV in conjunction with PET/CT imaging
  IV fluorine-18 labeled methylcholine before PET/CT: Intervention at pre-treatment, and at two timepoints post treatment intiation to determine Metabolically Active Tumor Volume (MATV) Response (30% or greater decline in MATV).
Period: Overall Study
Arm/Group | Received 18F-fluorocholine PET/CT
Started | 45
Completed | 42
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: 18F-fluoromethylcholine IV in conjunction with PET/CT imaging
  IV fluorine-18 labeled methylcholine before PET/CT: Intervention at pre-treatment, and at two timepoints post treatment intiation.
Arm/Group | Single Arm
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 42
Age, Continuous [Mean (Full Range); unit: Years] | 73 [70 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 42
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Metabolically Active Tumor Volume (MATV) Response
Description: Number of patients achieving 30% or greater reduction in MATV measured on 18F-fluorocholine PET/CT
Time Frame: 21 to 98 days
Measure: Count of Participants; unit: Participants
Arm/Group | Received 18F-fluorocholine PET/CT
Number analyzed (Participants) | 42
Participants | 20

2. Primary Outcome: Time to PSA Progression
Description: Time to PSA Progression between patients exhibiting MATV reduction greater or equal to 30% vs. MATV reduction less than 30%.
Time Frame: 2 years
Measure: Mean (Standard Error); unit: days
Arm/Group | Received 18F-fluorocholine PET/CT
Number analyzed (Participants) | 42
days
  MATV reduction > or = 30% | 194 (13.759)
  MATV reduction < 30% | 116 (26.929)

3. Primary Outcome: Proportional Hazards Regression Analysis of Time to PSA Progression
Description: PSA levels measured from the start of treatment over the period of follow-up were recorded. Time to PSA progression was calculated as the number of days from the start of treatment to the date of the first PSA test result that represented a 30% or greater increase from the PSA nadir, confirmed on the basis of repeated PSA measurements. For proportional hazards regression analysis, the percentage change in PSA level within 15 wk of starting treatment was calculated, using a 50% or greater decrease in PSA level as a predefined definition of PSA re- sponse based on Prostate Cancer Working Group guidelines.
Time Frame: Up to 15 week post-chemotherapy
Population: Twenty patients met the study criteria for an metabolically active tumor volume (MATV) response (30% or greater decline in MATV) response.
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Groups:
- Positive Metabolically Active Tumor Response: 18F-fluoromethylcholine IV in conjunction with PET/CT imaging
  IV fluorine-18 labeled methylcholine before PET/CT: Intervention at pre-treatment, and at two timepoints post treatment intiation. Positive Metabolically Active Tumor Volume (MATV) Response (30% or greater decline in MATV).
Arm/Group | Positive Metabolically Active Tumor Response
Number analyzed (Participants) | 42
Hazard Ratio | 0.246 [0.083 to 0.728]

ADVERSE EVENTS:
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 5/45
Other Adverse Events (participants affected / at risk) | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=45)
Severe Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Myocardial Ischemia, Diagnosis (Cardiac disorders) | 1 (1)
Severe Influenza (Infections and infestations) | 1 (1)
Obstructive Uropathy (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes